CLINICAL TRIAL: NCT07238062
Title: "An Intermediate Size Patient Population Expanded Access Protocol to Evaluate the Safety and Efficacy of Allogeneic HB-adMSCs for the Treatment of Multiple System Atrophy."
Brief Title: "An Intermediate Size Patient Population Expanded Access Protocol to Evaluate the Safety and Efficacy of Allogeneic HB-adMSCs (Hope Biosciences - Adipose Derived Mesenchymal Stem Cells) for the Treatment of Multiple System Atrophy."
Status: Temporarily not available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBMSA02
Record Dates: First submitted 2025-11-12; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Multiple System Atrophy
Keywords: msa; stem cells; MSCs
MeSH Terms: conditions — Multiple System Atrophy; Thyroid Dyshormonogenesis 2A

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: HB-adMSCs - Hope Biosciences Adipose Derived Mesenchymal Stem Cells — Intravenous and intrathecal infusion of Hope Biosciences autologous adipose-derived stem cells

SUMMARY:
This expanded access protocol is part of IND 32226 to evaluate efficacy and safety of multiple intravenous administrations of allogeneic HB-adMSCs for the treatment of Multiple System Atrophy for up to 7 adult patients who pass pre-screening and a completed screening. The subjects will receive 12 intravenous infusions of HB-adMSCs and 6 intrathecal injections of HB-adMSCs over the course of 44 weeks (1 infusion each month and 1 injection every other month).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 18-85 years of age
2. Participants must have a diagnosis of "Clinically Established" or "Clinically Probable" MSA.
3. Participants must have at least one brain MRI marker suggestive of MSA.
4. Participants must have both autonomic failure and either poorly L-dopa-responsive parkinsonism or cerebellar ataxia.
5. Female participants of childbearing potential should not be pregnant or plan to become pregnant during protocol participation and for 6 months after the last investigational product administration. Female participants of childbearing potential should confirm the use of one of the following contraceptive measures:

   * Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
   * Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
   * Barrier contraceptive methods (condoms, diaphragm, etc.).
   * Surgery (occlusion bilateral tubal ligation, hysterectomy, vasectomized partner).

   OR
   * Male participants if their sexual partners can become pregnant should ensure the use one of the following methods of contraception during protocol participation and for 6 months after the last administration of the investigated product:
   * Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
   * Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
   * Barrier contraceptive methods (condoms, diaphragm, etc.).
   * Surgery (vasectomy, occlusion bilateral tubal ligation (partner), hysterectomy (partner)).
6. Participants should be able to read, understand, and to provide voluntary consent.

Exclusion Criteria:

1. Women who are currently pregnant or lactating.
2. The participant has any active infection requiring medications per PI's discretion.
3. The participant has any clinical signs or symptoms of infection per PI's discretion.
4. The participant has hyperthermia or hypothermia.
5. The participant has any known recent (within the last 6 months) coagulation anomalies that are not being medically treated and are not stable per PI's discretion.
6. The participant has any abnormal laboratory values at the screening visit which the Investigator determines to be clinically significant and make the patient unsuitable for participation.
7. The Investigator determines the patient to be unsuitable for participation for other reasons, such as, but not limited to deep vein thrombosis (DVT), pulmonary embolus, cardiac arrhythmia, or those who have a prothrombotic condition, or who require persistent oxygen supplementation.
8. The participant has a substantial and persistent response to dopaminergic medications.
9. The participant has unexplained anosmia.
10. The participant has fluctuating cognition, early dementia, or hallucinations.
11. The participant has certain eye movement abnormalities.
12. The participant has any MRI findings that suggest an alternative diagnosis.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hope Biosciences Research Foundation, Sugar Land, Texas, United States

REFERENCES:
- See also: Hope Biosciences — http://www.hope.bio